CLINICAL TRIAL: NCT01220245
Title: Heparin-bonded Endoluminal Versus Surgical Femoropopliteal Bypass; a Multicentre Randomized Controlled Trial
Brief Title: SuperB Trial: SUrgical Versus PERcutaneous Bypass
Acronym: SuperB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Michel Reijnen, Principal Investigator, Rijnstate Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 721-070910
Record Dates: First submitted 2010-10-11; First posted 2010-10-13 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Cardiovascular Diseases
Keywords: endoluminal; surgical; bypass; patency; quality of life; multicentre; RCT; superficial femoral artery; vascular patency
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heparin-bonded endoluminal fempop bypass (Experimental): Heparin-bonded ePTFE endoluminal femoro-popliteal bypass versus surgical femoro-popliteal bypass
  Interventions: Procedure: Heparin-bonded ePTFE endoluminal fem-pop bypass
- Surgical femoro-popliteal bypass (Active Comparator): Surgical femoro-popliteal bypass.
  Interventions: Procedure: Surgical femoro-popliteal bypass.

INTERVENTIONS:
Procedure: Heparin-bonded ePTFE endoluminal fem-pop bypass — Heparin-bonded ePTFE endoluminal femoropopliteal bypass versus surgical femoropopliteal bypass
  Arms: Heparin-bonded endoluminal fempop bypass
Procedure: Surgical femoro-popliteal bypass. — Surgical femoro-popliteal bypass.
  Arms: Surgical femoro-popliteal bypass

SUMMARY:
In this multicentre Randomized Clinical Trial, the heparin-bonded endoluminal bypass will be compared to the surgical venous femoro-popliteal bypass, based on the non-inferiority principle for the patency. Besides equal patency, an improved quality of life is expected. Recruitment will take the first two years and patients will be followed during five years. Patients with an indication for surgical bypass, classified category 3-6 with a >50% stenosis or occlusion of the SFA over >/=10 cm in length will be included. At least one crural artery should be patent without significant lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Informed consent
* Novo stenosis, restenosis >50% or occlusion of the native SFA, all > 10cm in length
* Patent popliteal artery at the upper margin of the patella to the trifurcation
* Diameter native SFA and popliteal artery are 5.0-7.5 mm
* Indication for surgical bypass
* Distal run-off at least one crural artery without significant stenosis
* Ankle-brachial index (ABI) at rest < 0.8 in the study limb prior to procedure

Exclusion Criteria:

* Patient unsuitable for administration of contrast agent
* Pregnancy
* Dementia or altered mental status that would prohibit giving conscious informed consent
* Need for adjunctive major surgical or vascular procedures within one month
* Untreated flow-limiting aortoiliac occlusive disease
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment
* Femoral or popliteal aneurysm of target vessel
* Non-arthrotic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancies, dementia etc.) or other medical condition that would preclude compliance with study protocol
* Major distal amputation (above the transmetatarsal) in the study limb
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Known allergies to stent/stent-graft components
* History of prior life-threatening reaction to contrast agent
* Patients with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Planned surgical procedure or major amputation to occur after enrollment of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-10; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Primary (and -assisted) patency | 5 years
Quality of life | 5 years

SECONDARY OUTCOMES:
Secondary patency | 5 years
Complications | 5 years
Clinical improvement | 5 years
Re-intervention | 5 years
Target lesion revascularisation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MMJP Reijnen, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (6):
- Netherlands (6):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Slingeland Hospital, Doetinchem, Gelderland
  - Isala klinieken, Zwolle, Overijssel
  - Nij Smellinghe Hospital, Drachten, Provincie Friesland
  - Antonius Hospital, Sneek, Provincie Friesland
  - University Medical Centre Groningen, Groningen

REFERENCES:
- [Derived] van Walraven LA, Velandia-Sanchez A, Iqbal K, Zeebregts CJ, Holewijn S, Reijnen MMPJ. Impact on Hospital Resource Utilization of Endoluminal Bypass Using the Viabahn Endoprosthesis with Heparin Bioactive Surface Compared With Surgical Femoropopliteal Bypass. J Endovasc Ther. 2026 Feb;33(1):220-226. doi: 10.1177/15266028241245602. Epub 2024 Apr 9. PMID 38590283
- [Derived] Lensvelt MM, Holewijn S, Fritschy WM, Wikkeling OR, van Walraven LA, Wallis de Vries BM, Zeebregts CJ, Reijnen MM. SUrgical versus PERcutaneous Bypass: SUPERB-trial; Heparin-bonded endoluminal versus surgical femoro-popliteal bypass: study protocol for a randomized controlled trial. Trials. 2011 Jul 18;12:178. doi: 10.1186/1745-6215-12-178. PMID 21767371